CLINICAL TRIAL: NCT02107287
Title: Hypofractionated Intensity Modulated Radiation Therapy Plus Hormonal Therapy in Patients With High Risk Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sergio Faria (Other)
Responsible Party: Sponsor-Investigator, Sergio Faria, Associate Professor. Oncology., McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-519 GEN
Record Dates: First submitted 2012-08-22; First posted 2014-04-08 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: High Risk Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT Hypofractionated (Experimental): Neo-adjuvant hormone therapy for three months followed by IMRT combined with a 24-month hormonal therapy.
  Interventions: Radiation: IMRT Technique

INTERVENTIONS:
Radiation: IMRT Technique

SUMMARY:
Considering the promising results with hypofractionated in low and intermediate risk prostate cancer, our proposal is to translate this experience to patients with high risk prostate cancer. Patients with high risk disease would receive hypofractionated RT to the prostate and to the external and internal iliac lymph nodes using IMRT plus long-term hormonal therapy. The objective of the study is to show that long term grade>2 late toxicity is acceptable and similar to published data using hypofractionated technique in the prostate only.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven diagnosis of adenocarcinoma of the prostate meeting one of the following conditions:
* Clinical Stage >T3 or
* Gleason Score 8 or higher, or
* PSA level >20ng/ml
* Study entry PSA must be obtained within 6 weeks prior to protocol entry
* ECOG <2
* Age >18
* History and physical examination within 3 months
* Bone scan and CT scan of the abdomen and pelvis within 3 months with no evidence of bone metastases and no pelvic lymph nodes larger than 1.0cm, unless biopsy negative.
* CBC with differential within 6 weeks prior to protocol entry
* Absolute neutrophil count >2000cells/mm3
* Hemoglobin >8.0 g/dl (the use of transfusion to increase the Hg is acceptable)
* Testosterone level within 6 weeks of protocol entry
* Liver function tests
* Signed informed consent
* Prior use of hormonal therapy for prostate cancer is acceptable if less than 2 months.

Exclusion Criteria:

* Prior use of hormonal therapy for prostate cancer for more than 2 months. Previous use of finasteride or dutasteride is allowed.
* Prior invasive malignancy (except non-melanoma skin) unless disease-free for more than 5 years.
* Prior radiotherapy to the pelvis
* Life expectancy of less than 2 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Toxicity | First 3 months (acute toxicity)
  Acute and late toxicity following treatment with IMRT to the prostate and pelvic lymphatic chains will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (http://ctep.cancer.gov) for grading of all adverse events will be used in this study.

SECONDARY OUTCOMES:
Freedom from biochemical failure, patterns of failure. | At 5 years
  To measure freedom from biochemical failure (PSA measurement) at 5 years.

OTHER OUTCOMES:
Toxicity | 3 years
  Late effects will be also scored prospectively using the RTOG/EORTC late scoring system. Erectile dysfunction will be assessed by the SHIM questionnaire
Toxicity | 3 years
  Dose-volume histogram of the rectum and bladder will be correlated to the whole organ volumes doses and the development of GI and GU toxicity.
Rate of failure | 5 years
  To determine the rate of local, regional and distant failures.
Quality Assurance | 5 years
  To develop a quality assurance process for IMRT in prostate cancer at McGill University Health Center

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Faria, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada